CLINICAL TRIAL: NCT01024114
Title: Pilot Study to Evaluate the Incremental Diagnostic Value of a Combined Molecular Breast Imaging / Breast Tomosynthesis Modality
Brief Title: Study to Evaluate the Diagnostic Value of a Combined Molecular Breast Imaging/ Breast Tomosynthesis Modality
Status: Withdrawn | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amy L. Conners, MD, Mayo Clinic
Other Study IDs: 09-002678
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: MBI; Molecular Breast Imaging; Breast Cancer; Positive Molecular Breast Imaging scan.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Positive MBI scan: Women who are previously enrolled in an MBI study that present with a positive MBI scan.

SUMMARY:
The purpose of this pilot study is to investigate the potential clinical benefits of combining two new diagnostic tools to provide co-registered anatomical and functional information in the breast in patients with suspected breast cancer.

DETAILED DESCRIPTION:
The purpose of this pilot study is to obtain preliminary data on a new way of imaging the breast that combines the benefits of a 3-D anatomical technique (Digital Tomosynthesis) with those of a functional imaging technique (Molecular Breast Imaging). Combining data from these 2 modalities would provide co-registered functional and anatomical information on the breast, in the same way that PET/CT does today in oncology. This should greatly facilitate the evaluation and biopsy of lesions seen on MBI but occult on conventional mammography.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 25
* enrolled in one of the following protocols:

IRB # 08-005522: Evaluation of Molecular Breast Imaging in Patients with a High Likelihood of Ductal Carcinoma in Situ. 07-004241: Molecular Breast Imaging in the Preoperative Evaluation of Women with Biopsy Proven Breast Cancer. 1204-03: Evaluation of a Small Field of View Gamma Camera for Scintimammography in Patients with Atypical Ductal Hyperplasia, Atypical Lobular Hyperplasia, and Lobular Carcinoma In Situ. 07-003397: Comparison of MRI and Molecular Breast Imaging in Breast Diagnostic Evaluation. 17-05: Determination of the Sensitivity of a Dual-Headed Small Field of View Gamma Camera for the Detection of Small Breast Lesions.

* Digital mammogram at the Mayo Clinic within the past 30 days

Exclusion Criteria:

* They are unable to understand and sign the consent form
* They are pregnant or lactating
* They are physically unable to sit upright and still for 40 minutes.
* Recently enrolled on one of the ongoing tomosynthesis vs. mammography studies (rationale - avoid performing duplicate tomosynthesis studies in the same patient)

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will have had a molecular breast imaging study as part of their participation in one of the current research protocols evaluating this technology. A requirement for inclusion in this study is that patients will have had a digital mammography examination at Mayo Clinic within the past 30 days.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. O'Connor, Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic News — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0